CLINICAL TRIAL: NCT02920814
Title: Time Intensive Cognitive Behavioural Therapy for a Specific Phobia of Vomiting Using a Single Case Experimental Design
Brief Title: Time Intensive CBT for a Specific Phobia of Vomiting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/LO/0095
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2016-04

CONDITIONS: Specific Phobia of Vomiting; Emetophobia
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Time Intensive CBT for SPOV (Experimental): Time intensive CBT for SPOV involving 6 weekly sessions and 2 intensive days of 4 hours each (over 8 weeks in total).
  Interventions: Other: Cognitive Behavioural Therapy

INTERVENTIONS:
Other: Cognitive Behavioural Therapy — Time intensive CBT over 8 weeks, including 6 weekly sessions and two intensive days of 4 hours each.

SUMMARY:
The aims of this project are to determine the effectiveness of a time intensive form of Cognitive Behavioural Therapy (CBT) for Specific Phobia of Vomiting (SPOV). Current research shows that this brief format can be effective in other specific phobias e.g. insects and animals. However, to date limited research has been conducted on the effectiveness of time intensive forms of CBT for SPOV. A single case experimental design will be used to analyse specific and idiosyncratic outcome measures in 6-8 cases of SPOV, referred to the Centre for Anxiety Disorders and Trauma (CADAT) for treatment. Specifically, the project will explore the effectiveness of CBT delivered in a time-intensive format and imagery rescripting elements of the treatment. This initial study will provide important information about which elements of CBT are most effective at reducing targeted symptoms and whether symptom reduction can be achieved in a shorter number of sessions. It represents a crucial step before this format of CBT can be more rigorously evaluated and compared to other treatment approaches by Randomised Controlled Trial.

DETAILED DESCRIPTION:
Design A single case experimental design (ABACADA) will be used. A, B, C etc represents points of intervention and clinical contact with participants when standardised outcome measures will be administered by the treating clinician at each session. Phases A1, A2, A3 represent time between contact during which participants will undertake daily monitoring of idiosyncratic symptoms on Visual Analogue Scales (VAS) e.g. degree of avoidance, degree of worry, degree of nausea etc, so change between phases across time can be measured.

Participants will be randomly allocated to differing lengths of baseline phase (initial clinical assessment to first clinical session) with 4 potential arms (7, 10, 14, or 17 days). The first three clinical sessions (formulation, imagery rescripting and planning of intensive days) will take place weekly and last up to 1.5 hours. The two intensive days will last up to 4 hours each and take place shortly after the planning session and within a few days of each other. Three additional follow up sessions will be offered within 10 days of the intensive days (2 within one week, and the final session one week after). Follow up data will be collected by phone or post 3, 6 and 12 months post intervention.

Participants Participants will be recruited from consecutive referrals to CADAT for treatment of SPOV. Clients will have a diagnosis of SPOV as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) as their main presenting problem. They will be drawn from the CADAT waiting list, and if necessary from Improving Access to Psychological Therapy (IAPT) services at Southwark, Lambeth and Lewisham. These cases will be picked up by and treated at CADAT by qualified clinicians.

Participants are expected to be involved in the study for up to 8 weeks for the treatment phase, and 12 months for follow up data to be collected.

Recruitment Consultant Psychiatrist for the team at the Centre for Anxiety Disorders and Trauma will identify potential participants from the waiting list at CADAT who meet the inclusion criteria to take part in the study. Potential participants will then be asked if they would like to participate at the initial clinical assessment. They will be provided with an information sheet and the opportunity to ask questions before making a decision and giving informed consent.

Sample size It is estimated that 6-8 cases will be sufficient for a single case experimental design to demonstrate proof of concept. This is based on previous studies using a similar design.

Procedure Patients identified from the CADAT waiting list and who meet the study criteria will be asked at assessment if they would like to participate in the study. Those who are interested in taking part will be given an information sheet, and the opportunity to ask questions before making a decision on their participation. They will then be asked to provide informed written consent by signing a consent form before continuing with the study procedure. Clinicians will remind all participants of their right to withdraw from the study at any time, which will not affect their care or right to treatment as usual. Participants will then receive the time intensive form of CBT for their SPOV.

To ensure therapist adherence to the time intensive format of the treatment, a separate treatment protocol has been provided as part of Standard Operating Procedures. This protocol is as follows:

* Assessment and signing of consent form
* Session 1: Re-baseline & Formulation (including a conversation about early memory of vomiting)
* Session 2: Imagery Rescripting of early memory of vomiting
* Session 3: Planning for Intensive Days
* Intensive Day 1
* Intensive Day 2
* 3 short clinical follow up sessions

Standardised outcome measures will be collected at baseline, intervention and follow up phases. Participants will also be asked to collect daily idiosyncratic measures in between the intervention phases. Participants will be randomly allocated to differing lengths of baseline to the time of the intervention with 4 potential arms (7 days, 10 days 14 days or 17 days). This will be done using a simple spreadsheet by a Research Assistant at CADAT. The baseline discussion around the memory of vomiting, imagery re-scripting and treatment planning will consist of 1-1.5 hour sessions. Time intensive treatment will consist of two sessions over 2 days (4 hours each). Three additional follow up sessions will be administered, 2 within 1 week of the intensive days and a third 1 week after the second follow up session. The same standardised outcome measures will be collected at 3, 6 and 12 months by phone or post.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or over with a diagnosis of SPOV as defined by DSM-5
2. The individual describes the SPOV as their main psychological problem
3. The individual is able to read materials written in English and answer written questions
4. Individuals must have capacity to provide written informed consent

Exclusion Criteria:

1. Involvement in active CBT (imagery rescripting and/or exposure) within 2 years or inactive CBT within 1 year previous to this study
2. Individuals with a diagnosis of any other mental health disorder that required treatment in its own right
3. Individuals currently taking anti-anxiolytic medication where the dose has not been stable over one month prior to entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04; Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Specific Phobia of Vomiting Inventory (SPOVI) | 1 week
  A 14-item self-report measure that focuses on cognitive processes, safety seeking and avoidance behaviours (Veale et al, 2013). The total score ranges from 0 to 56. The scale has a two-factor structure, with one factor of 7 items characterized by avoidance (e.g. "I have been trying to avoid or control any thoughts or images about vomiting") and a second factor of 7 items comprised of threat monitoring (e.g. "I have been focused on whether I feel ill and could vomit rather than on my surroundings"). Cronbach's α is .91.

SECONDARY OUTCOMES:
Emetophobia Questionnaire | 1 week
  13-item self-report questionnaire that has good reliability and validity against a behavioural avoidance test (Boschen & Riddel, unpublished observations). The range is 13-65. The EmetQ has 3 factors. Factor 1 had 6 items focused on avoidance of travel, movement, or locations. Factor II was comprised of 3 items, which centred on themes of dangerousness of exposure to vomit stimuli. Factor III consisted of 4 items that focus on avoidance of others who may vomit. Cronbach's α is 0.82.
Patient Health Questionnaire (PHQ-9) | 1 week
  9-item measure of depressive symptoms, based on DSM-IV. The total score ranges from 0 to 27 and Cronbach's α was .86.
Generalised Anxiety Disorder (GAD7) | 1 week
  7-item scale and is designed to measure the severity of symptoms of generalized anxiety disorder. The total score ranges from 0 to 21 and the Cronbach's α was 0.92.
Work and Social Adjustment Scale | 1 week
  5 item scale that is designed to measure interference in life.
IAPT Employment Status Questions | 1 week
  Questions relating to current employment status, Statutory Sick Pay and benefits.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Anxiety Disorders and Trauma, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No